CLINICAL TRIAL: NCT01266590
Title: Effect of LY2216684 on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Study of LY2216684 and Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12600; H9P-EW-LNCK (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 + digoxin (Experimental): Two oral 0.5-milligrams (mg) (two 0.25-mg tablets) doses of digoxin separated by 12 hours on Day 1, followed by once daily 0.25-mg (single 0.25-mg tablet) dose of digoxin on Days 2-14. Daily oral 18-mg (two 9-mg tablets) doses of LY2216684 on Days 8-14.
  Interventions: Drug: LY2216684; Drug: Digoxin

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Digoxin — Administered orally

SUMMARY:
The purpose of this study is to determine how much digoxin gets into the blood stream and how long it takes the body to get rid of it when given with LY2216684. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or Women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] greater than (>) 40 milli-International Units/milliliter (mIU/mL).
* Have a body weight >50 kilograms (kg).
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator (potassium, magnesium, and calcium values must be within the normal range).
* Have normal renal function defined as an estimated creatinine clearance of at least 80 milliliters/minute (mL/min) as calculated with the Cockcroft-Gault equation.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, digoxin, or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of significant dysrhythmias or atrioventricular (AV) block.
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication (including hormonal contraceptives) within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor, except for influenza vaccinations.
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of P-glycoprotein (P-gp) and Cytochrome (P45) (CYP) within 30 days prior to dosing.
* Have donated blood of more than 500 milliliters (mL) within the last month.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to check-in until completion of the study (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participant unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2216684 + Digoxin
Started | 30
Completed | 24
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | LY2216684 + Digoxin
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Digoxin: Maximum Plasma Concentration (Cmax)
Description: Cmax of digoxin when administered alone and when co-administered with LY2216684.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 7 and 14
Population: All participants who received at least 1 dose of study drug and had evaluable Cmax values.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms/milliliter (ng/mL)
Groups:
- Digoxin: 0.5-milligrams (mg) (two 0.25-mg tablets) digoxin administered orally twice on Day 1 and 0.25-mg (single 0.25-mg tablet) digoxin administered orally once daily on Days 2 through 7.
- LY2216684 + Digoxin: 0.25-mg (single 0.25-mg tablet) digoxin and 18-mg (two 9-mg tablets) LY2216684 administered orally once daily on Days 8 through 14.
Arm/Group | Digoxin | LY2216684 + Digoxin
Number analyzed (Participants) | 27 | 25
nanograms/milliliter (ng/mL) | 1.433 [1.266 to 1.622] | 1.424 [1.254 to 1.617]

2. Primary Outcome: Pharmacokinetics of Digoxin: Time to Maximum Plasma Concentration (Tmax)
Description: Tmax of digoxin when administered alone and when co-administered with LY2216684.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 7 and 14
Population: All participants who received at least 1 dose of study drug and had evaluable Tmax values.
Measure: Median (Full Range); unit: hours
Arm/Group | Digoxin | LY2216684 + Digoxin
Number analyzed (Participants) | 25 | 25
hours | 2.00 [0.50 to 3.00] | 1.00 [0.50 to 4.00]
Statistical Analysis 1: Comparison: Digoxin vs LY2216684 + Digoxin; Test type: Superiority or Other; p = 0.0664, Wilcoxon Signed Rank

3. Primary Outcome: Pharmacokinetics of Digoxin: Area Under the Concentration Time Curve at Steady State Over the Dosing Interval (AUCt)
Description: AUCt at steady state of digoxin when administered alone and when co-administered with LY2216684.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose on Days 7 and 14
Population: All participants who received at least 1 dose of study drug and evaluable AUCt values.
Measure: Geometric Mean (90% Confidence Interval); unit: hours*nanograms/milliliter (h*ng/mL)
Arm/Group | Digoxin | LY2216684 + Digoxin
Number analyzed (Participants) | 27 | 25
hours*nanograms/milliliter (h*ng/mL) | 14.6 [13.2 to 16.1] | 14.3 [12.9 to 15.8]

ADVERSE EVENTS:
Groups:
- Digoxin 0.5mg: 0.5-milligrams (mg) (two 0.25-mg tablets) digoxin administered orally twice on Day 1.
- Digoxin 0.25mg: 0.25-mg (single 0.25-mg tablet) digoxin administered orally once daily on Days 2 through 7.
Arm/Group | Digoxin 0.5mg | Digoxin 0.25mg | LY2216684 + Digoxin
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 3/30 | 4/28 | 16/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Digoxin 0.5mg (N=30) | Digoxin 0.25mg (N=28) | LY2216684 + Digoxin (N=27)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram pr shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Semenuria (Renal and urinary disorders) | 0/18 (0) | 0/17 (0) | 2/16 (3)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Genital disorder male (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 1/16 (1)
Penile size reduced (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 1/16 (1)
Testicular disorder (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 1/16 (1)
Testicular pain (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 2/16 (2)
Testicular swelling (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 1/16 (1)
Testis discomfort (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 1/16 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days